CLINICAL TRIAL: NCT00615069
Title: A Clinical Study Evaluating the Use of the GORE EXCLUDER® AAA Endoprosthesis - 31mm In the Primary Treatment of Infrarenal Abdominal Aortic Aneurysms
Brief Title: Study of the Large Diameter GORE EXCLUDER® AAA Endoprosthesis in Abdominal Aneurysms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA 03-02
Record Dates: First submitted 2007-12-20; First posted 2008-02-14 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 31 mm GORE EXCLUDER® Test Subjects (Experimental): GORE EXCLUDER® AAA Endoprosthesis - 31 mm device implanted for the primary treatment of infrarenal abdominal aortic aneurysms (AAA)
  Interventions: Device: 31 mm GORE EXCLUDER® AAA Endoprosthesis

INTERVENTIONS:
Device: 31 mm GORE EXCLUDER® AAA Endoprosthesis — GORE EXCLUDER® AAA Endoprosthesis - 31 mm device implanted for the primary treatment of infrarenal abdominal aortic aneurysms (AAA)
  Other Names: GORE EXCLUDER® Bifurcated Endoprosthesis

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the 31 mm GORE EXCLUDER® AAA Endoprosthesis in the treatment of infrarenal abdominal aortic aneurysms

DETAILED DESCRIPTION:
The primary objective of this study was to estimate the safety of the 31 mm GORE EXCLUDER® AAA Endoprosthesis as compared to open surgical repair when used in the treatment of infrarenal abdominal aortic aneurysms. A secondary objective was to compare device performance of the original GORE EXCLUDER® AAA Endoprosthesis to the 31mm EXCLUDER when used in the treatment of infrarenal abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Infrarenal AAA > or equal to 4.5 cm in diameter
* Proximal infrarenal aortic neck length > or equal 15mm
* Anatomy meets 31mm EXCLUDER specification criteria
* Access vessel able to receive 20 Fr. introducer sheath
* Life expectancy >2 years
* Surgical candidate
* ASA Class I, II, III, or IV
* NYHA Class I, II, III
* 21 years of age or older
* Male or infertile female
* Ability to comply with protocol requirements including follow-up
* Signed Informed Consent Form

Exclusion Criteria:

* Mycotic or ruptured aneurysm
* Participating in another investigational device or drug study within 1 year
* Documented history of drug abuse within 6 months
* Coexisting thoracic aortic aneurysm (50% larger than proximal aorta)
* Myocardial infarction or cerebral vascular accident within 6 weeks
* Pulmonary insufficiency requiring chronic home oxygen therapy or inability to ambulate due to pulmonary function
* Renal insufficiency (Creatinine > 2.5 mg/dL) without dialysis
* Iliac anatomy that would require occlusion of both internal iliac arteries
* "Planned" occlusion or reimplantation of significant mesenteric or renal arteries
* "Planned" concomitant surgical procedure or previous major surgery within 30 days
* Previous prosthesis placement in the same position of the aorta or iliac arteries
* Degenerative connective tissue disease, e.g., Marfans and Ehlers Danlos Syndrome
* Proximal neck angulation > 60 degrees
* Presence of significant thrombus at arterial implantation sites

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon S Matsumura, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- St. Vincent Healthcare, Billings, Montana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: May 2006 - Mar 2009 (Study Subjects and Continued Access)
Groups:
- 31 mm GORE EXCLUDER® Test Subjects: GORE EXCLUDER® AAA Endoprosthesis - 31 mm device implanted for the primary treatment of infrarenal abdominal aortic aneurysms (AAA). This study was designed for primary analysis following one year of follow up, however, total subject follow up is 5 years post treatment. Participant Flow results reflect the final (5 year) data.
Period: Overall Study
Arm/Group | 31 mm GORE EXCLUDER® Test Subjects
Started | 35
Completed | 19
Not Completed | 16
Not completed — Death | 10
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- 31 mm GORE EXCLUDER® Test Subjects: GORE EXCLUDER® AAA Endoprosthesis - 31 mm device implanted for the primary treatment of infrarenal abdominal aortic aneurysms (AAA). This study was designed for primary analysis following one year of follow up, however, total subject follow up is 5 years post treatment.
Arm/Group | 31 mm GORE EXCLUDER® Test Subjects
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Time to First Major Adverse Event Experienced by Subjects From the Time of Treatment Through 1 Year
Time Frame: Treatment through 1 year post-procedure (365 days)
Measure: Mean (Standard Error); unit: days
Groups:
- 31 mm GORE EXCLUDER® Test Subjects: GORE EXCLUDER® AAA Endoprosthesis - 31 mm device implanted for the primary treatment of infrarenal abdominal aortic aneurysms (AAA). This study was designed for primary analysis following one year of follow up.
Arm/Group | 31 mm GORE EXCLUDER® Test Subjects
Number analyzed (Participants) | 35
days | 84.0 (24.2)
Statistical Analysis 1: Comparison: 31 mm GORE EXCLUDER® Test Subjects; Log-rank test of freedom from major adverse events through 1 year, 31 mm GORE EXCLUDER® Test Subjects vs historical open surgical control Subjects; Test type: Superiority or Other; p = 0.003, Log Rank

2. Secondary Outcome: Number of Subjects With One or More of the Following Events: Type I Endoleak, Device Migration, Major Procedural Bleeding Complications
Time Frame: Treatment through 1 year window post-procedure (through end of 1 year window, 546 days)
Measure: Number; unit: Participants
Arm/Group | 31 mm GORE EXCLUDER® Test Subjects
Number analyzed (Participants) | 35
Participants | 4
Statistical Analysis 1: Comparison: 31 mm GORE EXCLUDER® Test Subjects; Estimation of Hazard ratio of the 31 mm GORE EXCLUDER® Test Subjects vs original GORE EXCLUDER® AAA Endoprosthesis Subjects (original PMA subjects) using Cox Regression, not a powered analysis; Test type: Superiority or Other; Hazard Ratio (HR) = 1.241, 95% CI 2-sided [0.428 to 3.603]

ADVERSE EVENTS:
Time Frame: Adverse Event results reflect the final (through 5 year) data.
Description: Note: only major/minor classification was collected. All events classified as 'Major' are in 'Serious adverse events', 'Minor' events are in 'Other adverse events'. Major adverse events had to result in: a)therapy and short hospitalization b)major therapy/increase in level of care/prolonged hospitalization c)permanent adverse sequelae or d)death.
Arm/Group | 31 mm GORE EXCLUDER® Test Subjects
Serious Adverse Events (participants affected / at risk) | 24/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 31 mm GORE EXCLUDER® Test Subjects (N=35)
Bleeding (Blood and lymphatic system disorders) | 3
Cardiac (Cardiac disorders) | 7
Bowel (Gastrointestinal disorders) | 7
Endoleak (General disorders) | 2
Other (General disorders) | 7
Sepsis (Infections and infestations) | 2
Wound (Injury, poisoning and procedural complications) | 4
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Neurologic (Nervous system disorders) | 7
Renal Function (Renal and urinary disorders) | 2
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 6
Lumen Obstruction (Vascular disorders) | 1
Vascular (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 31 mm GORE EXCLUDER® Test Subjects (N=35)
Bleeding (Blood and lymphatic system disorders) | 6
Cardiac (Cardiac disorders) | 9
Bowel (Gastrointestinal disorders) | 6
Endoleak (General disorders) | 18
Other (General disorders) | 16
Other Device Complication (General disorders) | 2
Wound (Injury, poisoning and procedural complications) | 8
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neurologic (Nervous system disorders) | 5
Genitourinary (Renal and urinary disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 6
Vascular (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator willpostpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating study sites.